CLINICAL TRIAL: NCT05946954
Title: Evaluation of Soft and Hard Tissue Changes Following Immediate Implant Using Immediate Dentoalveolar Restoration Versus Ice Cream Cone Technique In Cases With Labial Plate Dehiscence: A 1-Year Randomized Clinical Trial
Brief Title: Immediate Implant Placement Using Immediate Dentoalveolar Restoration Versus Ice Cream Cone Technique With Labial Plate Dehiscence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aya Sharaf (Other)
Responsible Party: Sponsor-Investigator, Aya Sharaf, Dentist, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2623
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Immediate Implant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group Immediate Dentoalveolar Restoration (Experimental): * After applying anesthesia to the maxillary tuberosity, a full thickness crestal incision was made following the distal contour of the maxillary right second molar. This incision was followed by a palatal release incision to access the donor area.
  * The flap was raised in the tuberosity area Then, the bone graft was harvested from the underlying bone by using a 1 cm wide flat chisel and a surgical hammer.
  * The corticocancellous graft was manipulated using a rongeur to reproduce the shape of the peri-implant bone defect.
  * The graft was carefully inserted to the level of the implant platform Finally, a screw-retained resin provisional crown, relined over a polyetheretherketone (PEEK) anti-rotation abutment, was placed out of occlusion, establishing the ideal emergence profile to accommodate the soft tissues and to promote a thicker and more stable gingival tissue margin
  Interventions: Procedure: Immediate Dentoalveolar Restoration
- Control group Ice cream cone technique (Active Comparator): Ice cream cone technique
  1. Resorbable collagen membrane will be cut confirming to the size and shape of the defect of labial bone plate dehiscence. The membrane will be placed against internal surface of the extraction socket against the remaining buccal plate of bone.
  2. The gap between the collagen membrane and the implant fixture will be filled with xenograft particulates.
  The membrane will be folded in palatal direction to seal the socket in an ice cream cone shape, then will be secured using resorbable sutures to prevent dislodgment of the blood clot and bone grafting material
  Interventions: Procedure: Ice cream cone technique

INTERVENTIONS:
Procedure: Immediate Dentoalveolar Restoration — Topical anesthesia will be administered using an infiltration technique. • Atraumatic extraction will be done with the aid of periotome and Luxators. • The extraction socket will be debrided to remove any residual debris or granulation tissue. •. Socket walls will be checked using a periodontal probe to ensure integrity of all sockets walls except the labial bone plate which must show a dehiscence.
  • Implant placement will be done according to manufactures' instructions; drills will be used sequentially in a more palatal direction leaving a buccal jumping gap of at least 2mm. All implants will engage at least 3 mm apical to the apical end of the socket with adequate primary stability
  Arms: Intervention group Immediate Dentoalveolar Restoration
Procedure: Ice cream cone technique — Topical anesthesia will be administered using an infiltration technique. • Atraumatic extraction will be done with the aid of periotome and Luxators. • The extraction socket will be debrided to remove any residual debris or granulation tissue. •. Socket walls will be checked using a periodontal probe to ensure integrity of all sockets walls except the labial bone plate which must show a dehiscence.
  • Implant placement will be done according to manufactures' instructions; drills will be used sequentially in a more palatal direction leaving a buccal jumping gap of at least 2mm. All implants will engage at least 3 mm apical to the apical end of the socket with adequate primary stability
  Arms: Control group Ice cream cone technique

SUMMARY:
: Evaluation of Soft and Hard Tissue Changes following Immediate Implant using Immediate Dentoalveolar Restoration Versus Ice Cream Cone technique for management of Cases With Labial Plate Dehiscence

DETAILED DESCRIPTION:
In patients with labial plate dehiscence in the esthetic zone, there is no difference between the use of Immediate Dentoalveolar Restoration Versus Ice Cream Cone technique in conjunction with immediate implant placement in enhancing the amount of bone labial to the implant

ELIGIBILITY:
Inclusion Criteria:

* Non-restorable teeth in the esthetic zone with a defect of labial bone.
* Teeth with no acute inflammation.
* Patients are free from any systemic condition that may affect the healing.
* Availability of bone apical and palatal to the socket to provide primary stability
* Good oral health.
* Willingness to sign the informed consent form.

Exclusion Criteria:

Heavy smoker (> 10 cigarettes/day)

* Pregnant females
* Contraindication for Implant surgery.
* Patients with poor oral hygiene.
* Acute inflammation in the site of implantation and adjacent tissue.
* A history of radiotherapy in the head or neck region.
* Patients with systemic diseases like uncontrolled diabetes mellitus, coagulation disorders, alcohol or drug abuse not suitable for implantation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Bucco/facial-palatal ridge thickness | 1 year
  Impressions were taken with addition silicone before tooth extraction, after six months of implant placement (immediately after the placement of the definite crown) and 12 months after crown installation. Casts were then obtained with special gypsum stone type IV.Casts were measured by a dentist not involved in the study with a digital caliper. Three reference points were measured from the free gingival margin to the apex at the implant site and in the contralateral tooth: 1 mm, 3 mm and 6 mm

SECONDARY OUTCOMES:
Radiographic bucco-palatal bone changes | 1 year
  The bucco-palatal width of the alveolar bone will be measured perpendicular to the long axis of the alveolar bone; the 3 measurements will be the coronal width (CW), middle width (MW), and apical width (AW). Each measurement will be recorded at different times
3. Radiographic width of bone labial to the implant | 1 year
  Amount of bone labial to the implant will be measured perpendicular to the vertical line of the implant surface at the implant neck level or the top of the buccal bone (which is regarded as 0 mm), 3 mm and 6 mm apical to the implant neck Each measurement will be recorded at different times (at day 0 after finishing the procedure, 6 and 12 months post-operatively)
Radiographic vertical bone changes | 1 year
  Vertical bone height will be measured. Measurement will be taken at highest point of the remaining labial/buccal plate of bone using the implant neck as a reference point. Each measurement will be recorded at different times and the difference between pre and post-operative measurements will be determined as the gain in labial/buccal vertical bone dimension
Esthetic evaluation (The pink esthetic score) | 1 year
  The pink esthetic score will be calculated on the parameters defined by (Fürhauser et al. 2005). Clinical photographs will be taken to evaluate peri-implant soft tissue through evaluating seven variables compared to a natural reference tooth including: mesial papilla, distal papilla, soft-tissue level, soft-tissue contour, alveolar process deficiency, soft- tissue color and texture. Using a 0-1-2 scoring system, 0 being the lowest, 2 being the highest value. The maximum achievable PES is 14.
Implant stability | 6 months
  implant stability will be measured using Ostell which has a scale ranges from 1 to 100, the higher the ISQ the more stability
Gingival Thickness | 1 year
  Gingival thickness will be evaluated 2 mm below the gingival margin with a short needle for and silicon disk stop. The needle will be inserted perpendicular to the mucosal surface, through the soft tissues with light pressure until a hard surface was reached. The silicone disc stop was then mounted in close contact with the gingival tissue surface. The insertion depth was assessed with a digital caliper accurate to the nearest 0.1 mm
Width of the Keratinized Tissue | 1 year
  It will be evaluated from the gingival margin to the mucogingival junction (MGJ). The MGJ was assessed with roll technique
Midfacial recession | 1 year
  Corono-apical distance between the peri-implant soft tissue margin and the cemento-enamel junction (CEJ) of the homologous contralateral tooth
Post-Operative Pain | 7 days
  Pain will be assessed post-surgically using the Visual Analogue Scale (VAS) with numbers from 0 to 10 score zero represented no pain while score 10 represented the worst pain imaginable
Post-Operative patient's Satisfaction | 1 year
  Three Yes or No Questions will be asked to the patient about his overall satisfaction about the procedure
Post-operative swelling | 7 days
  Swelling will be assessed post-surgically using the Verbal Rating Scale (VRS) (García et al. 2008):
  * Absent (no swelling),
  * Slight (intraoral swelling at the operated area),
  * Moderate (moderate intraoral swelling at the operated area) and
  * Intense (intensive extraoral swelling extending beyond the operated area)

IPD SHARING:
Plan to Share IPD: Undecided